CLINICAL TRIAL: NCT06147648
Title: Prospective, Multicenter Clinical Study of Prolonged-release Tacrolimus in Stable Liver Transplant Recipients
Brief Title: Early Conversion of Prolonged-release Tacrolimus in Liver Transplantation.
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Principal Investigator, QIAN LU, professor, Beijing Tsinghua Chang Gung Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 23163-4-01
Record Dates: First submitted 2023-10-12; First posted 2023-11-27 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Liver Transplantation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Single arm observational registry study Drug: Tacrolimus Sustained-release Capsules (Experimental): Drug: Tacrolimus Sustained-release Capsules
  After liver transplantation, immediate-release tacrolimus was administered for acute rejection prevention, and after 3 months, it was converted into tacrolimus sustained-release capsules in a ratio of 1:1 to 1:1.2; (The specific medication plan is decided by the clinician according to the actual situation)
  Interventions: Drug: Tacrolimus Sustained-release Capsules

INTERVENTIONS:
Drug: Tacrolimus Sustained-release Capsules — Transition from Immediate-release tacrolimus to prolonged-release tacrolimus at 3 months after liver transplantation

SUMMARY:
Tacrolimus is a commonly used immunosuppressant after liver transplantation. A once-daily administration of prolonged-release tacrolimus has been found to improve patient compliance and offer good efficacy and safety. Moreover, there is evidence that this prolonged-release formulation mitigates renal impairment and metabolic syndrome in transplant recipients. Foreign studies have confirmed that it is safe and feasible for liver transplant recipients to switch from immediate-release tacrolimus to prolonged-release tacrolimus during the stable period. At the same time, patients with early conversion are more likely to benefit in terms of graft survival and renal function recovery, and the proportion of drug conversion needs to be further explored.

This study aims to assess the efficacy and safety of switching from immediate-release tacrolimus to prolonged-release tacrolimus three months after liver transplantation. Furthermore, it seeks to investigate the impact of this conversion on indicators such as liver function, kidney function, metabolic disease incidence, and infection incidence in patients.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old and above
2. 3 months after liver transplantation;
3. Stable use of immediate-release tacrolimus for at least one month before enrollment in the study;
4. The serum levels of aspartate aminotransferase [AST] and alanine aminotransferase [ALT] were within the normal range; ….

Exclusion Criteria

1. Multi-organ combined transplantation or multiple liver transplantation;
2. Multiple organ recipients or those who have previously transplanted any organs；
3. Adjuvant liver transplantation or use of bioartificial liver therapy;
4. Prior to joining the group, they had received treatment with immune checkpoint (ICIs);
5. Participation in any other clinical study within 3 months prior to enrollment;
6. Use of tacrolimus sustained release capsules before enrollment;
7. Tacrolimus trough concentration lower than 5 ng/ml at the time of screening;
8. Acute rejection occurred within one month prior to enrollment; ….

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2025-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of biopsy-confirmed acute rejection (BPAR) within 3, 6, and 12 months after conversion | within 3, 6, and 12 months after conversion

SECONDARY OUTCOMES:
Graft survival rate and patient survival rate at 12 months after conversion | 12 months after conversion
The conversion dose ratio from ordinary tacrolimus to tacrolimus sustained-release capsules; | 3 months after liver transplantation
Incidence of infection (viral, bacterial and fungal) at 12 months after conversion; | 12 months after conversion;
Observe the serum aspartate aminotransferase (AST) levels of subjects at 3, 6, and 12 months after switching to the prolonged-release tacrolimus. | within 3,6,12 months after conversion
Observe the serum alanine aminotransferase (ALT) levels of subjects at 3, 6, and 12 months after switching to the prolonged-release tacrolimus. | within 3,6,12 months after conversion
Observe the creatinine clearance rate of subjects at 3, 6, and 12 months after switching to the prolonged-release tacrolimus. | within 3,6,12 months after conversion